CLINICAL TRIAL: NCT00307853
Title: A Randomised, Double - Blind, Placebo Controlled Clinical Trial to Assess the Efficacy of the Homeopathic Medication TRAUMEEL S in Controlling Pain After Total Knee and Total Hip Arthroplasty.
Brief Title: TRAUMEEL for Pain After Total Knee/Hip Arthroplasty
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of patients
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Menachem Oberbaum, MD, Shaare Zedek Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP 06
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Total Knee and Total Hip Arthroplasty
Keywords: homeopathy; pain; traumeel s; total knee arthroplasty; total hip arthroplasty
MeSH Terms: conditions — Pain | interventions — Traumeel S

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): TraumeelS
  Interventions: Drug: Traumeel S; Other: Traumeel S
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Traumeel S — All patients will receive an intra-operative injection of either Traumeel S or placebo solution. Afterwards, verum or indistinguishable placebo tablets, PO, two tablets five times daily from day 0 to 6 post-operatively, and two tablets three times daily from day 7 until day 21. To the extent possible, administration of tablets should be equally spaced between morning and evening (e.g. every 6 hours) at the same time every day.
  Arms: 1
Other: Traumeel S — All patients will receive an intra-operative injection of either Traumeel S or placebo solution. Afterwards, verum or indistinguishable placebo tablets, PO, two tablets five times daily from day 0 to 6 post-operatively, and two tablets three times daily from day 7 until day 21. To the extent possible, administration of tablets should be equally spaced between morning and evening (e.g. every 6 hours) at the same time every day.
  Arms: 1
Other: Placebo — All patients will receive an intra-operative injection of either Traumeel S or placebo solution. Afterwards, verum or indistinguishable placebo tablets, PO, two tablets five times daily from day 0 to 6 post-operatively, and two tablets three times daily from day 7 until day 21. To the extent possible, administration of tablets should be equally spaced between morning and evening (e.g. every 6 hours) at the same time every day.
  Arms: Placebo

SUMMARY:
We hypothesize that Traumeel S is more effective than placebo in reducing 48-hour mean cumulative morphine consumption following Total Knee or Hip Arthroplasty.

224 patients, meeting all inclusion and none of exclusion criteria, will be enrolled in the trial. Patients will be randomized to receive either intraoperative injection and post operative oral Traumeel S Tablets or placebo injection (normal saline) and indistinguishable oral placebo tablets. Baseline measurements of relevant outcome measures will taken preoperatively.

In the recovery room, the patient will begin to receive IV Dipyrone (Optalgin) 1000mg, for a total of 4 doses during the first 24 hours postoperatively (1000 mg every 6 hours). Once back in the ward, the patient will be connected to an IV Patient-Controlled Analgesia (PCA) device, enabling the self-administration of morphine at a set dose of 1mg every 8 minutes, should the patient require it. The PCA memory registers the time and dose, and the data will be used later to evaluate post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex undergoing unilateral THAP or TKAP.
* Age over 18 years.
* Signature upon informed consent form

Exclusion Criteria:

* Participation in another clinical trial within 4 weeks prior to enrollment.
* Refused to give verbal consent to the telephone interviews
* Impossibility to be reached during the 14-17 days post operative
* Inability to comply with the study protocol for any other reason
* Previous major surgical procedure on ipsilateral leg.
* Current use of analgesics for any other reason.
* A history of chronic pain syndrome.
* Abused legal or illicit drug use.
* Hypersensitivity to botanicals of the Compositae family
* Known sensitivity to paracetamol, codeine or tramadol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative 48-hour postoperative morphine consumption as consumed by the patient via the PCA device | 48h

SECONDARY OUTCOMES:
AUC of NRS scores for days 14-17. | 14-17d
Cumulative 24-hour postoperative morphine consumption as consumed by the patient via the PCA device | 24h
Number of primary oral analgesic tablets ingested between days 14-17 | 14-17d
ESR and hs-CPR at three and six days and six weeks | 6d and 3weeks
IL-6 at three and six days | 3 and 6d
Post operative blood loss | postoperative period
WOMAC | 6 weeks
Safety of post operative treatment | 6 weeks
Development of acute confusional state in the postoperative period | 14-17d

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (2):
- Israel (2):
  - Dept. of Orthopedic Surgery, Shaare Zedek Medical Center, Jerusalem
  - Department of Orthopedics, Meir Medical Center, Kfar Saba